CLINICAL TRIAL: NCT01898364
Title: An Open-label, Multicenter, Multinational, Ascending Dose Study of the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Exploratory Efficacy of Repeated Biweekly Infusions of neoGAA in naïve and Alglucosidase Alfa Treated Late-onset Pompe Disease Patients.
Brief Title: Safety and Efficacy Evaluation of Repeat neoGAA Dosing in Late Onset Pompe Disease Patients.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDR12857; 2012-004167-42 (EudraCT Number); U1111-1144-7725 (Other: (UTN))
Record Dates: First submitted 2013-07-02; First posted 2013-07-12 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Pompe Disease; Glycogen Storage Disease Type II (GSD II); Acid Maltase Deficiency
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- GZ402666 (neoGAA) Group 1 - 5 mg (Experimental): Intravenous infusion of 5mg neoGAA to treatment naïve late onset Pompe disease patients once every other week for a total of 24 weeks
  Interventions: Drug: GZ402666
- GZ402666 (neoGAA) Group 1 - 10 mg (Experimental): Intravenous infusion of 10mg neoGAA to treatment naïve late onset Pompe disease patients once every other week for a total of 24 weeks.
  Interventions: Drug: GZ402666
- GZ402666 (neoGAA) Group 1 - 20 mg (Experimental): Intravenous infusion of 20mg neoGAA to treatment naïve late onset Pompe disease patients once every other week for a total of 24 weeks.
  Interventions: Drug: GZ402666
- GZ402666 (neoGAA) Group 2 - 5 mg (Experimental): Intravenous infusion of 5mg neoGAA once every other week for a total of 24 weeks to late onset Pompe disease patients previously treated with alglucoside alfa.
  Interventions: Drug: GZ402666
- GZ402666 (neoGAA) Group 2 - 10 mg (Experimental): Intravenous infusion of 10mg neoGAA once every other week for a total of 24 weeks to late onset Pompe disease patients previously treated with alglucoside alfa.
  Interventions: Drug: GZ402666
- GZ402666 (neoGAA) Group 2 - 20 mg (Experimental): Intravenous infusion of 20mg neoGAA once every other week for a total of 24 weeks to late onset Pompe disease patients previously treated with alglucoside alfa.
  Interventions: Drug: GZ402666

INTERVENTIONS:
Drug: GZ402666 — Pharmaceutical form:lyophilized powder reconstituted for infusion Route of administration: intravenous

SUMMARY:
Primary Objective:

To evaluate the safety and tolerability of neoGAA in treatment naïve and alglucosidase alfa treated late-onset Pompe disease patients.

Secondary Objective:

To evaluate the pharmacokinetics, pharmacodynamics of neoGAA in treatment naïve and alglucosidase alfa treated late-onset Pompe disease patients.

To evaluate the effect of neoGAA on exploratory efficacy endpoints in treatment naïve and alglucosidase alfa treated late-onset Pompe disease patients.

DETAILED DESCRIPTION:
Screening: within 90 days Period of treatment: 24 weeks (including 13 bi-weekly infusions) Post treatment evaluation visit: 2 weeks after last neoGAA infusion (at Week 27) End of study visit: 4 weeks after last neoGAA infusion (at Week 29) Total duration: approximately 41 weeks

ELIGIBILITY:
Inclusion criteria :

For both Group 1 and Group 2:

* Male or female patients with confirmed acid α-glucosidase (GAA) enzyme deficiency from any tissue source and/or confirmed GAA gene mutation and without known cardiac hypertrophy.
* Patient willing and able to provide signed informed consent
* Patient is able to ambulate 50 meters (approximately 160 feet) without stopping and without an assistive device. Use of assistive device for community ambulation is appropriate.
* Patient has a forced vital capacity (FVC) in upright position of ≥50% predicted.
* The patient, if female and of childbearing potential, must have a negative pregnancy test [urine beta-human chorionic gonadotropin (β-hCG)] at baseline.

Group 2 patients only:

- The patient has been previously treated with alglucosidase alfa for at least 9 months.

Exclusion criteria:

For both Group 1 and Group 2:

* Patient is wheelchair dependent.
* Patient requires invasive-ventilation (non-invasive ventilation is allowed).
* Patient is participating in another clinical study using investigational treatment.
* Patient, in the opinion of the Investigator, is unable to adhere to the requirements of the study.
* Patient has clinically significant organic disease (with the exception of symptoms relating to Pompe disease), including clinically significant cardiovascular, hepatic, pulmonary, neurologic, or renal disease, or other medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, precludes participation in the study or potentially decreases survival.
* Patient cannot submit to MRI examination because of a formal contraindication such as a pacemaker, implanted ferromagnetic metals, anxiety disorder, etc.

Group 1 only:

- Patient has had previous treatment with alglucosidase alfa or any other enzyme replacement therapy (ERT) for Pompe disease.

Group 2 only:

- Patient has a high risk for a severe allergic reaction to neoGAA (i.e. previous moderate to severe anaphylactic reaction to alglucosidase alfa and/or patient has immunoglobulin (Ig) E antibodies to alglucosidase alfa, and/or a history of sustained high immunoglobulin G (IgG) antibody titers to alglucosidase alfa that in the opinion of the investigator suggest a high risk for an allergic reaction to neoGAA).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-08-19 (Actual); Primary Completion 2015-02-25 (Actual); Study Completion 2015-02-25 (Actual)

PRIMARY OUTCOMES:
Adverse events | screening/baseline to Week 25
Laboratory assessments including hematology, biochemistry and urinalysis | screening/baseline to Week 25
Vital signs | screening/baseline to Week 25

SECONDARY OUTCOMES:
Electrocardiogram | screening/baseline, Week 1, Week 13, Week 25
Immunogenicity assessments | screening/baseline to Week 29
Cmax | Week 1, Week 13, Week 25
AUC | Week 1, Week 13, Week 25
t1/2 | Week 1, Week 13, Week 25
Skeletal muscle glycogen content | screening/baseline, Week 27
Skeletal muscle magnetic resonance images for qualitative and quantitative muscle degenerative assessments. | screening/baseline, Week 27
Urinary Hex4 | screening/baseline to Week 25
Functional assessments including 6 Minute Walk Test (6MWT) | screening/baseline, Week 13, Week 25
  Functional Assessment includes - pulmonary function testing (PFT) endpoints, Gait, Stair, Gower's Maneuver, Chair (GSGC), Gross Motor Function Measure-88 (GMFM-88), Quick Motor Function Test (QMFT), hand-held dynamometer testing, Pediatric Quality of Life Inventory Multidimensional Fatigue Scale (PedsQL)
Quality of life assessments | screening/baseline, Week 13, Week 25

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (17):
- United States (7):
  - Investigational Site Number 840006, Phoenix, Arizona
  - Investigational Site Number 840010, Jacksonville, Florida
  - Investigational Site Number 840001, Kansas City, Kansas
  - Investigational Site Number 840008, St Louis, Missouri
  - Investigational Site Number 840002, Durham, North Carolina
  - Investigational Site Number 840009, Dallas, Texas
  - Investigational Site Number 840003, Fairfax, Virginia
- Investigational Site Number 056001, Leuven, Belgium
- Investigational Site Number 208001, København Ø, Denmark
- France (3):
  - Investigational Site Number 250001, Marseille
  - Investigational Site Number 250003, Nice
  - Investigational Site Number 250002, Paris
- Germany (3):
  - Investigational Site Number 276003, Mainz
  - Investigational Site Number 276001, München
  - Investigational Site Number 276002, Münster
- Investigational Site Number 528001, Rotterdam, Netherlands
- Investigational Site Number 826003, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Derived] Dimachkie MM, Barohn RJ, Byrne B, Goker-Alpan O, Kishnani PS, Ladha S, Laforet P, Mengel KE, Pena LDM, Sacconi S, Straub V, Trivedi J, Van Damme P, van der Ploeg AT, Vissing J, Young P, Haack KA, Foster M, Gilbert JM, Miossec P, Vitse O, Zhou T, Schoser B; NEO-EXT investigators. Long-term Safety and Efficacy of Avalglucosidase Alfa in Patients With Late-Onset Pompe Disease. Neurology. 2022 Aug 1;99(5):e536-e548. doi: 10.1212/WNL.0000000000200746. PMID 35618441